CLINICAL TRIAL: NCT02095210
Title: Phase 1 Study, Evaluating HER2 PET Imaging in Breast Cancer Patients Using [68GA]ABY-025
Brief Title: HER2 PET Imaging in Breast Cancer Patients Using [68GA]ABY-025
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: Dorte Nielsen (Other)
Responsible Party: Sponsor-Investigator, Dorte Nielsen, Professor, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MA1021
Record Dates: First submitted 2011-05-31; First posted 2014-03-24 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: HER2-positive Breast Cancer
Keywords: PET scan; HER2; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 68Ga-ABY-025; Product Labeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- [68Ga]ABY-025 PET imaging (Experimental): Radiolabeled [68Ga]ABY-025
  Interventions: Other: Radiolabeled [68Ga]ABY-025

INTERVENTIONS:
Other: Radiolabeled [68Ga]ABY-025 — Single dose of 100 μg ABY-025 labeled with 500 MBq gallium-68, administrated as a slow intravenous injection. All patients will receive the same dose.
  Other Names: tracer for HER2

SUMMARY:
This is an open-labeled, exploratory, single center study. Patients with a big primary breast cancer (≥ 3 cm) or metastatic first line, routinely have their HER2-expression determined by biopsy. Patients having a HER2-positive tumor will be recruited to the study. A [18F]FDG PET/ceCT scan is performed for the measurement of uptake in the tumour and diagnosis of possible metastases. Each subject will receive a single injection of the investigational product [68Ga]ABY-025, followed by measurement of uptake in the tumour or metastases and in normal organs. The investigations will be repeated after HER2 directed therapy.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

1. Subject is > 18 years of age
2. Histologically or cytologically confirmed diagnosis of breast adenocarcinoma ≥ 3 cm determined by ultrasound, or locally advanced breast cancer (LABC: T3-4NxMx or TxN2-3Mx)
3. HER2-positiv breast cancer first recurrence
4. HER2-positiv breast cancer primary metastatic
5. HER2 status has been determined on biopsy material from the primary tumour and found to be HER2-positive, defined as a DAKO HercepTest™ score of 3+ or else 2+ and FISH positive
6. [18F]FDG PET/ceCT performed within 7 days before administration of IMP
7. ECOG performance status of =< 2
8. Hematological, liver and renal function test results within the following limits:

   * White blood cell count: > 2.0 x 10^9/L
   * Haemoglobin: > 5.0 mmol/L
   * Platelets: > 50.0 x 10^9/L
   * ALT, ALP: =< 3 times Upper Limit of Normal
   * Bilirubin =< 2.0 times Upper Limit of Normal
   * Serum creatinine: Within Normal Limits
9. A negative pregnancy test (serum beta-HCG) at screening for all subjects of childbearing potential
10. Subject is capable to undergo the diagnostic investigations to be performed in the study
11. Informed consent

Exclusion Criteria:

* 1. Known hypersensitivity to Dotarem® 2. Active known autoimmune disease or history of autoimmune disease 3. Active serious infection according to investigator evaluation 4. Known HIV positive or chronically active hepatitis B or C 5. Administration of other investigational medicinal product within 30 days of screening 6. Pregnant or breast-feeding 7. Women capable of childbearing not using a sufficient non-hormonal method of birth control 8. Other primary malignancies (including primary brain tumors) within the last 5 years before inclusion, with exception of sufficiently treated in situ carcinoma of the cervix, squamous carcinoma of the skin or sufficiently controlled limited basal cell carcinoma of the skin 9. Signs of any other disease, metabolic or psychological dysfunction, findings at physical examination or laboratory findings, which give reasonable suspicion of a disease or condition that would contraindicate use of the IMP, could influence the patient's compliance with the study routines or involves an increased risk for treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2014-08-13 (Actual); Study Completion 2014-08-13 (Actual)

PRIMARY OUTCOMES:
to evaluate the uptake distribution of the HER2-binding imaging agent [68Ga]ABY-025 by PET imaging in breast cancer patients with biopsy-identified HER2 expression | 28 days from last dose of study drug

SECONDARY OUTCOMES:
Assess concordance of [68Ga]ABY-025 uptake with [18F]FDG PET uptake before and after HER2 therapy | within 14 days before study drug
2. pharmacokinetics of [68Ga]ABY-025 and whole-body dosimetry of [68Ga]ABY-025 | 6 weeks after last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata K Tuxen, MD, P.hd., Principal Investigator — Consultant
Locations (1):
- Herlev University Hospital, Oncology Department, Herlev, Denmark